CLINICAL TRIAL: NCT05945381
Title: Evaluation of Efficiency, Acceptance and the Durability of Glass-Ionomer Sealing Technique on Hypersensitive MIH (Molar Incisor Hypomineralisation) Teeth With and Without Enamel Breakdown - a Cohort Study
Brief Title: Effect of Glass-Ionomer Sealing Technique on Hypersensitive Teeth With Molar Incisor Hypomineralisation
Acronym: MIH_GIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB 047/23
Record Dates: First submitted 2023-06-06; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Hypersensitive; Molar Incisor Hypomineralization; Pit and Fissure Sealants
MeSH Terms: conditions — Hypersensitivity; Molar Hypomineralization; Van der Woude syndrome

STUDY DESIGN:
Intervention Model Description: The tooth will be cleaned with a prophylactic paste and brush for complete debris and plaque removal. The tooth will then be dried with a cotton roll, as the patient doesn't tolerate the air-drying (which is the case in SCASS 2 and 3). Moisture control will be kept with cotton roll, the tooth is then sealed with a hard setting glass-ionomer cement (IonoStar Plus, VOCO, Germany) followed by an application of a surface coat (Easy Glaze, VOCO, Germany) for moisture and dehydration protection after sealant application. The distributed questionnaire will include questions regarding the attitude of the child's caregiver to the idea and their estimation of the child's fair regarding dental visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GIC on MIH (Experimental): see below
  Interventions: Combination Product: GIC on MIH

INTERVENTIONS:
Combination Product: GIC on MIH — Subjects will be seated in a dental chair set-up using standard infection control guidelines. Then the study and its objectives will be explained to the patients and their caregivers. The tooth will be cleaned with a prophylactic paste and brush for complete debris and plaque removal. The tooth will then be dried with a cotton roll, as the patient doesn't tolerate the air-drying (which is the case in SCASS 2 and 3). Moisture control will be kept with cotton roll, the tooth is then sealed with a hard setting glass-ionomer cement (IonoStar Plus, VOCO, Germany) followed by an application of a surface coat (Easy Glaze, VOCO, Germany) for moisture and dehydration protection after sealant application. The distributed questionnaire will include questions regarding the attitude of the child's caregiver to the idea and their estimation of the child's fair regarding dental visit.

SUMMARY:
This single armed cohort study is aimed to assess the acceptance, durability and efficiency of glass-Ionomer sealing technique on hypersensitive MIH molars (TNI-3 & 4a/b/c) clinically shortly (15 minutes) after the application and after a time period of 3 months.

DETAILED DESCRIPTION:
The main assumption of the study is that sealing of hypersensitive MIH molars (TNI-3 & 4a/b/c) using glass-ionomer cement reduces the degree of hypersensitivity after direct placement and within a period of time. Moreover, glass-ionomer sealing has a good durability in hypomineralized teeth and is known to be acceptable due to it's easy and fast application.

The aim of this study is to assess the change in the degree of hypersensitivity in the sealed MIH (molar incisor hypomineralisation) tooth / teeth (IonoStar Plus, VOCO-Germany) in the same visit (15 Minutes after the application) and in the 3 months' recall-visit according to Schiff Cold Air Sensitivity (SCASS) Test and the self-report of the patient using Wong- Baker Faces Rating Scale.

This single armed cohort study will be undertaken at the Department of Preventive and Pediatric Dentistry at the University of Greifswald from approximately May 2023 to Autumn 2024. After assessment of eligibility and informed consent for participation in the study, hypersensitivity of the affected MIH permanent molars will be assessed using air blast before the treatment using SCASS (Schiff cold air sensitivity Scale) and VAS (Visual analogue scale) in order to record the degree of sensitivity and pain perception of the child. After initial assessment, the affected teeth are prepared to receive a Glass- Ionomer cement fissure sealant (IonoStar Plus, VOCO GmbH Germany).

The level of tooth sensitivity will be assessed again 15 minutes after the treatment and in the regular 3 months follow up via air blast test (Schiff Cold Air Sensitivity Scale), the pain perception is being recorded with VAS (Visual analogue scale) by an independent observer, dental assistant and the operating dentist. The independent observer will assess the cooperation and behaviour of the child throughout the treatment using FBRS (Frankl behavioural rating scale) and FIS (Facial image scale).

The durability of the fissure sealant will be assessed using the modified USPHS criteria in the 3 months' follow-up. After the dental visit, the participating child the accompanying parent or caregiver, the dental operator receives a short questionnaire to be filled out.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported hypersensitive MIH molar (MIH-TNI 3 & 4a/b/c).
* Children & adolescents without systematic health diseases.
* No sealing therapy or application of desensitizing agent on the MIH-teeth within 1 month before participation in the study.
* Agreement to voluntary participation in the study.

Exclusion Criteria:

* Patients with acute pain/ patients with signs or symptoms to be treated.
* Patients with systemic disease that require special attention during their dental treatment.
* Parents / children who refused to participate in the study. - MIH teeth with signs of irreversible pulpitis.
* Allergy against any ingredients of the material.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity (mid-term) | 3 months
  Change in the degree of hypersensitivity in the sealed MIH tooth / teeth (IonoStar Plus, VOCO-Germany) in the 3 months' recall-visit according to Schiff Cold Air Sensitivity (SCASS) Test. (scale: 0;1;2;3; max hypersensitivity: 3; no hypersensitivity 0)
Hypersensitivity (short-term) | 15 minutes
  Change in the degree of hypersensitivity in the sealed MIH tooth / teeth (IonoStar Plus, VOCO-Germany) after 15 minutes according to Schiff Cold Air Sensitivity (SCASS) Test. (scale: 0;1;2;3; max hypersensitivity: 3; no hypersensitivity 0)

SECONDARY OUTCOMES:
child acceptance of procedure | 15 minutes
  - Assessment of acceptance of the child toward the procedure using Likert Scale (scale: 1-5)
hypersensitivity: assessment of the child | 15 minutes
  Change in the degree of hypersensitivity in the sealed MIH tooth / teeth (IonoStar Plus, VOCO-Germany) regarding self-report of the patient using Wong- Baker Faces Rating Scale. (0-10; 0=no hurt; 10=hurts worst)
durability | 3 months
  Evaluation of durability of the sealant material on the MIH-teeth using modified USPHS assessment's criteria (in 3 months' recall).
  Scale Alpha: No loss of sealing material Bravo: Partial loss of sealing material Charlie: Loss of restorative material

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Splieth, Prof., Study Director — Dep. preventive & pediatric dentistry, University of Greifswald
Locations (1):
- Department of Preventive and Pediatric Dentistry, University of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No